CLINICAL TRIAL: NCT02388581
Title: Multicentre, Prospective Study of First-line Antibiotic Therapy for Early-stage H. Pylori-Positive Gastric Pure (de Novo) Diffuse Large B-cell Lymphoma and Potential Predicting Factor for Treatment Outcome
Brief Title: First-line Antibiotic Therapy for Early-stage HP(+) Gastric Pure DLBCL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Health Research Institutes, Taiwan (Other)
Collaborators: National Taiwan University Hospital (Other); Mackay Memorial Hospital (Other); China Medical University Hospital (Other); Taichung Veterans General Hospital (Other); Changhua Christian Hospital (Other); National Cheng-Kung University Hospital (Other); Chang Gung Memorial Hospital (Other); Kaohsiung Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T2214
Record Dates: First submitted 2014-12-04; First posted 2015-03-17 (Estimated); Last update posted 2016-03-25 (Estimated); Status verified 2015-12

CONDITIONS: Gastric Diffuse Large B-cell Lymphoma
Keywords: Helicobactor pylori, Hp; mucosa-associated lymphoid tissue-type lymphoma, MALToma
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone | interventions — Lansoprazole; Amoxicillin; Clarithromycin; Metronidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Anti-H. pylori Therapy (Experimental): Lansoprazole, Amoxicillin, Clarithromycin, Metronidazole
  Interventions: Drug: Lansoprazole, Amoxicillin, Clarithromycin, Metronidazole

INTERVENTIONS:
Drug: Lansoprazole, Amoxicillin, Clarithromycin, Metronidazole — Anti-H. pylori Therapy
  Other Names: Anti-H. pylori Therapy

SUMMARY:
Aims: A nationwide study to prospectively validate

1. The complete histological and molecular remission rate for antibiotics as 1st-line therapy for early-stage Hp-positive gastric pure (de novo) DLBCL
2. The durability of complete histological remission after antibiotics
3. The usefulness of pattern of NF-kB, BCL10, BAFF, and CagA by IHC staining in prospectively predicting the Hp-dependence of gastric pure (de novo) DLBCL
4. The frequency of t(11;18)(q21;q21) translocation in gastric pure (de novo) DLBCL in Taiwan.
5. The association between the CYP2C18/CYP2C19 genetic polymorphisms and eradication of Hp infection after antibiotics.

DETAILED DESCRIPTION:
The study will validate the use of antibiotics as first-line therapy for stage IE (and perhaps IIE-1) Hp-positive gastric pure (de novo) DLBCL. The status of NF-kB, BCL10, BAFF, and CagA IHC nuclear staining will help to tailoring the treatment for early-stage gastric pure (de novo) DLBCL. And 50-60% of stage IE / IIE-1 pure (de novo) DLBCL patients can be cured by 2-weeks of antibiotics rather than the 6-months of relatively toxic front-line systemic chemotherapy. The investigators shall also elucidate the distribution of CYP2C18/19 in patients with pure (de novo) DLBCL and their association with the efficacy of sequential antibiotics for eradication of Hp infection.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically confirmed H. pylori-positive primary gastric pure (de novo) gastric DLBCL.
2. Patient must have no prior chemotherapy or radiotherapy for his/her gastric pure (de novo) gastric DLBCL.
3. Patients must have evaluable disease by endoscopy and/or by computed tomography.
4. Patients must have documented H. pylori infection before treatment, if any of the following test show positive result: histology, rapid urease test (CLO-test), C13 urease breath test, and serology.
5. Patients must have either stage IE or IIE-1 disease, according to an adaptation of the Ann Arbor staging system modified by Musshoff for primary extranodal lymphoma.
6. Patients who are either newly diagnosed or already starting anti-H. pylori therapy but not have follow-up endoscopy and biopsy are eligible.
7. Patient must have signed the informed consent, and agree to provide achieved pathologic material for immunohistochemical / fluorescence in situ hybridization study and RT-PCR for t(11;18)(q21;q21) determination.

Exclusion Criteria:

1. Patients with extensive gastrointestinal tract involvement.
2. Patients with previous history of extranodal lymphoma.
3. Patients with stage IIE-2 or beyond disease: infiltration of regional lymph node.
4. Patients with cardiopulmonary status that do not allow repeat endoscopy.
5. Patients with prior chemotherapy or radiotherapy for their primary gastric lymphoma.
6. Patients who had previous anti-H. pylori therapy and without pretreatment pathology achieve material for histological review and immunohistochemical study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-12; Primary Completion 2017-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
The pathologic complete remission rate (%) for antibiotics as 1st-line therapy for early-stage Hp-positive gastric pure (de novo) DLBCL | 10 years
The median time to pathologic complete remission (months) after completion of antibiotics for Hp-dependent gastric pure (de novo) DLBCL (patients have pCR after Hp eradication therapy [antibiotics]) | 10 years
The relapse-free survival of early-stage Hp-positive gastric pure (de novo) DLBCL who received antibiotics as 1st-line therapy | 10 years
  A nationwide study to prospectively validate

SECONDARY OUTCOMES:
The overall survival of early-stage Hp-positive gastric pure (de novo) DLBCL who received antibiotics as 1st-line therapy | 10 years
The Hp eradication rate (%) | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Sung-Hsin Kuo, MD, PhD., Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Health Research Institutes, Zhunan, Miaoli County, Taiwan